CLINICAL TRIAL: NCT00573001
Title: Phase 3 Randomized Trial Evaluating the Virological Efficacy and the Tolerance of 4 New Simplified Antiretroviral Treatments in Naive HIV-1 Infected Patients in Dakar and Yaounde
Brief Title: Evaluation of 4 New Simplified Antiretroviral Treatments in Naive HIV-1 Infected Patients in Africa (ANRS 12115 DAYANA)
Acronym: DAYANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other); Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS12115 DAYANA; IMEA 032
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: naive; HIV-1; simplified treatment; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Nevirapine; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Tenofovir/Emtricitabine (Truvada) and Nevirapine
- 2 (Experimental)
  Interventions: Drug: Tenofovir (Viread) and Lopinavir/Ritonavir (Aluvia)
- 3 (Experimental)
  Interventions: Drug: Tenofovir/Emtricitabine (Truvada) and Zidovudine
- 4 (Active Comparator)
  Interventions: Drug: Tenofovir/Emtricitabine/Efavirenz (Atripla)

INTERVENTIONS:
Drug: Tenofovir/Emtricitabine (Truvada) and Nevirapine — Tenofovir/Emtricitabine(Truvada) 245/200mg 1cp/day ; Nevirapine 200mg 2cp/day after first 14 days
  Other Names: Truvada
  Arms: 1
Drug: Tenofovir/Emtricitabine/Efavirenz (Atripla) — Tenofovir/Emtricitabine/Efavirenz (Atripla) 300/200/600mg 1cp/day
  Other Names: Atripla
  Arms: 4
Drug: Tenofovir (Viread) and Lopinavir/Ritonavir (Aluvia) — Tenofovir (Viread) 300mg 1cp/day ; Lopinavir/Ritonavir (Aluvia) 400/100mg 4cp/day
  Other Names: Viread; Aluvia
  Arms: 2
Drug: Tenofovir/Emtricitabine (Truvada) and Zidovudine — Tenofovir/Emtricitabine (Truvada) 245/200mg 1cp/day ; Zidovudine 300mg 2cp/day
  Other Names: Truvada
  Arms: 3

SUMMARY:
The goal of this trial is to demonstrate that new treatments are as effective as a reference triple-agent regimen in driving plasma viral load below the detection limit early during treatment (16 weeks). These simplified treatments involve fewer tablets and intakes, fixed-dose combinations, and also radically new strategies such as boosted protease inhibitor and tenofovir.

DETAILED DESCRIPTION:
The efficacy of antiretroviral treatments in sub-Saharan Africa has been demonstrated in cohort studies and pilot trials. The treatment regimens tested in these studies were derived from those used in pre-marketing trials conducted in industrialized countries.

However, the choice of antiretrovirals for national programs in poor countries is largely based on drug availability through the Access program, together with cost and supply considerations, rather than on field evaluations of recommended strategies.

Concomitantly with the development of antiretroviral access programs in the southern hemisphere, first-line treatments in industrialized countries have tended to become simpler, thereby improving their convenience and reducing the incidence and severity of their adverse effects. These simplified treatments involve fewer tablets and intakes, fixed-dose combinations, and also radically new strategies such as boosted protease inhibitor and tenofovir. These simplified strategies are being extensively evaluated in industrialized countries.

Long-term economic benefits will be a determining factor in the adoption of these strategies by poor countries.

Methods:

We will conduct a phase-III unblinded randomised trial focusing on the early virologic efficacy, tolerability and immuno-virologic efficacy of four simplified antiretroviral regimens given for 96 weeks to previously untreated HIV-1-infected patients in Senegal and Cameroon. The following four simplified treatments will be tested: TDF/FTC/NVP, LPV/TDF, TDF/FTC/AZT and TDF/FTC/EFV. The required number of patients (n=120) is compatible with the short-term recruitment capacity of two clinical investigation centers in Senegal and Cameroon.

Objective:

The goal of this trial is to demonstrate that these new treatments are as effective as a reference triple-agent regimen (TDF/FTC/EFV) in driving plasma viral load below the detection limit early during treatment. The principal objective is to identify simplified treatments capable of driving viral load below 50 copies/mL at week 16 in at least 50% of patients. If successful, the initial treatments will be continued and re-assessed at 96 weeks.

Study design:

120 patients previously unexposed to antiretroviral drugs will be recruited over a one-year period in two treatment centers in Dakar (Infectious Diseases department of Fann University Hospital) and Cameroon (Yaounde Military Hospital and Principal Hospital)

Expected results:

This study is fully in keeping with WHO/UNAIDS recommendations on antiretroviral treatment simplification in poor countries. These new treatments must be evaluated in the countries concerned, given the often very advanced stage of HIV disease at diagnosis, intercurrent health disorders, and local socioeconomic conditions.

This trial is not designed to compare these new treatments with one another, but rather to select the most promising treatments for future use. These preliminary results will help with the choice of treatment strategies for cohort studies and large-scale randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years for Senegal and over 21 years for Cameroon
* HIV-1 infected patient
* patient naive from any antiretroviral treatment
* CD4 cell count over 50 cells per mm3
* contraceptive method use
* informed consent signed

Exclusion Criteria:

* opportunistic infection ongoing or any other serious pathology
* ongoing treatment with rifampicine
* severe renal or hepatic impairment
* HbSAg positive
* Hemoglobine under 8g/L
* Neutrophils under 500 cells per mm3
* ongoing pregnancy or breastfeeding
* treatment by contra-indicated drugs (as described in study drugs notices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with viral load below 50 copies/mL | week 16

SECONDARY OUTCOMES:
Percentage of patients with viral Load under 50 copies/ml and under 400 copies/ml | W4, W12, W24, W36, W72, and W96
Severe adverse event onset, metabolic alterations, lipodystrophia | J0, W16, W24, W48, W72, W96
Residual ARV plasmatic concentration | W4, W48
CD4 count evolution | J0, W4, W16, W24, W36, W48, W72, W96
quality of life parameters, observance | J0, W4, W8, W12, W16, W24, W36, W48, W72, W96

CONTACTS AND LOCATIONS:
Overall Officials: Landman Roland, MD, Principal Investigator — Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba; Sow Papa Salif, MD, Principal Investigator — Hopital de Fann, Dakar; Koulla Shiro Sinata, MD, Principal Investigator — Hopital Central Yaoundé
Locations (2):
- Hopital Central, Yaoundé, Cameroon
- Hopital de Fann, Dakar, Senegal

REFERENCES:
- See also: Sponsor web page — http://www.anrs.fr